CLINICAL TRIAL: NCT01374698
Title: Preprocedural Asprin Reload for Native Coronary Disease Treated by Angioplasty: Reperfusion Indexes Evaluation and Improvement of Clinical Outcome -PANTAREI Study
Brief Title: Aspirin Reload Before Percutaneous Coronary Intervention: Reperfusion Indexes Evaluation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Violi, Prof., University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sapienza
Record Dates: First submitted 2011-05-06; First posted 2011-06-16 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Arteriosclerosis
Keywords: PCI; Aspirin; Reload
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Active Comparator): All patients who meet the eligibility criteria will be randomized in a 1:1 manner to receive, before the coronary percutaneous procedure, an oral aspirin reload (325 mg)or placebo.
  Interventions: Drug: Aspirin
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Drug: Aspirin — Aspirin 325 mg
  Arms: Aspirin

SUMMARY:
This is a prospective, randomized study conducted in patients undergoing coronary revascularization procedures (PCI) through angioplasty. All patients who meet the eligibility criteria will be randomized to receive, before the procedure, an oral aspirin reload (325 mg) and to be re-evaluated at 60 minutes, 120 minutes, 6 hours, 48 hours, 5 and 30 day, 3 and 6 months.

DETAILED DESCRIPTION:
Study population will be composed of 60 patients with a native coronary chronic occlusion with a vessel diameter equal or superior to 3 mm. The vessels must be treated through a balloon angioplasty and must be completely covered with two stent maximum with a maximum length ≤ 33 mm each. The native coronary chronic occlusion is defined as a native coronary obstruction, if established from at least 30 days, without lumen continuity and a "Thrombolysis In Myocardial Infarction" (TIMI) flow grade equal or superior to 1.

Patient must be treated with an chronic (at least 7 days) oral 100 mg/die aspirin treatment. After the eligibility criteria confirmation, the patient will be randomized with a 1:1 ratio to receive the aspirin reload or not.

Coronary angiographies will be evaluated by the centralized laboratory with the Coronary Quantitative Angiography method.

Myocardial necrosis indexes, ejection fraction, TIMI frame count (TFC) and myocardial blush grade (MBG) variations will represent the short term primary end-points. Clinical events incidence, including death, myocardial infarction, target vessel revascularization and stent thrombosis, will be evaluated at 1, 6 and 12 months.

Study design In every patient will be performed a baseline blood sample collection to evaluate inflammation, platelet activation and oxidative stress indexes. After baseline collection of blood samples, computer-generated random sequence were used for randomization to an oral aspirin reload administration or not.

Every patient, as guidelines described, will receive an oral clopidogrel reload (300 mg) that will be turned to 75 mg/die oral administration for the next 6 months. After procedure, the patient will turn back to the chronic aspirin 100 mg/die oral treatment.

After a percutaneous access will be obtained, it will be administered a 5000 U unfractioned heparin bolus, treating the dose to obtain a clotting time equal or superior to 250 seconds during the intervention.

A basal angiography will be performed in at least two orthogonal adjoining projections using a diagnostic 6F catheter. Every angiograms must include at least 2 cm catheter length to allow accurate quantitative coronary angiographic evaluations.

Target lesion will be crossed by a 0,0014" metallic guide and a single proper-dimensions-balloon predilatation will be performed inflating a nominal pression to the balloon for 15 seconds long.

In 1 minute from the dilatation will be implanted a sirolimus eluting stent (SES; Cypher ™, Cordis, Johnson& Johnson). Stent deployment will be obtained by an high pressure 10 seconds balloon inflate (more than 15 atm) without any second dilatation. No direct stent implantation will be realized.

TFC and MBG will be evaluated before and after the procedure. At 60 and 120 minutes and at 6 hours after the procedure a blood sample collection will be performed to evaluate the same baseline indexes. After 48 hours, 5 and 30 day ejection fraction will be re-evaluated. Every 3 months, for 12 months at least, patient will receive an ambulatorial follow up to recognize the new ischemic symptoms or instrumental signs onset.

Statistical Considerations Previous observations reported that after revascularization procedure has been observed a 35% plasmatic thromboxane levels increase (in vivo platelet activation index) in patients receiving chronic aspirin treatment (7 days). Hypothesizing that the oral aspirin reload could produce a 25% absolute reduction in plasmatic thromboxane levels (10%) this study needs a 50 patients for every treatment arm sample size (1-beta=90%; alfa=5%).

ELIGIBILITY:
Inclusion Criteria:

* De novo native coronary chronic occlusion with a reference diameter equal or superior to 3 mm programmed treatment;
* 100 mg/die oral aspirin treatment for at least 7 days before the procedure;
* Target lesion must be covered with two stent maximum with a maximum length ≤ 33 mm each
* Signed written informed consent

Exclusion Criteria:

* Aspirin, bisulphate clopidogrel, ticlopidine, heparin, contrast agent or heavy metals known allergy that cannot been medically handled;
* Target occlusion localized inside a previously implanted graft
* Target occlusion localized inside a vessel segment previously underwent stent-positioning
* Target occlusion localized inside a vessel with other occlusion not-to-be treated with the target occlusion same stent(s)
* Target occlusion localized inside a vessel with other occlusions need to be treated with balloon angioplasty
* Other techniques than balloon angioplasty target occlusion pre-treatment such as atherectomy, laser intervention or thrombectomy
* Coronary brachytherapy treated patients
* Ejection fraction equal or minor to 30%
* Renal insufficiency (creatinine >3.0 mg/dl)
* Warfarin-treated patients
* Life expectancy minor to 12 months
* Heart transplanted patients
* Patients still enrolled in some other study, both pharmacological both not

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of pre procedural aspirin overload effect on markers of platelet activation after percutaneous coronary intervention (PCI) | Change from baseline at 120 minutes
  Changes from the baseline of platelet activation markers (thromboxane) after 60, 120 minutes and 6 hours from the end of percutaneous coronary intervention.

SECONDARY OUTCOMES:
Reperfusion Index | At the end of the procedure (an expected average of 30 minutes)
  Changes of TFC and MBG (used to assess myocardial perfusion) before and after PCI.
Myocardial damage assessed by mean peak values of cardiac troponin I (cTnI) after the percutaneous coronary procedure. | Changes from baseline at 6 hours
  At 60 and 120 minutes and at 6 hours after the procedure a blood sample collection will be performed to evaluate Myocardial necrosis indexes.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Basili, MD, Principal Investigator — Sapienza-Univerity of Rome; Violi Francesco, Prof., Study Chair — Sapienza; Gaetano Tanzilli, Prof., Principal Investigator — Sapienza; Marcello Dominici, MD, Principal Investigator — Division of Cardiology, Department of Interventional Cardiology, Santa Maria University Hospital, Terni, Italy
Locations (1):
- Sapienza University of Rome, Rome, Italy

REFERENCES:
- [Derived] Basili S, Tanzilli G, Raparelli V, Calvieri C, Pignatelli P, Carnevale R, Dominici M, Placanica A, Arrivi A, Farcomeni A, Barilla F, Mangieri E, Violi F. Aspirin reload before elective percutaneous coronary intervention: impact on serum thromboxane b2 and myocardial reperfusion indexes. Circ Cardiovasc Interv. 2014 Aug;7(4):577-84. doi: 10.1161/CIRCINTERVENTIONS.113.001197. Epub 2014 Jul 29. PMID 25074252